CLINICAL TRIAL: NCT01173536
Title: A Multiple-Dose, Randomized, Double-Blind, Placebo-Controlled, Active-Comparator, Parallel-Group Study to Investigate the Effect of GDC-0449 on the QT/QTc Interval in Healthy Female Subjects
Brief Title: A Study to Investigate the Effect of GDC-0449 on the QT/QTc Interval in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHH4871g
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — HhAntag691; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: moxifloxacin; Drug: placebo
- B (Active Comparator)
  Interventions: Drug: moxifloxacin; Drug: placebo
- C (Experimental)
  Interventions: Drug: GDC-0449; Drug: placebo

INTERVENTIONS:
Drug: GDC-0449 — Oral repeating dose
  Arms: C
Drug: moxifloxacin — Oral single dose
  Arms: A; B
Drug: placebo — Oral repeating dose

SUMMARY:
This is a Phase I, single-center, three-arm, randomized, double-blind, active- and placebo-controlled study to investigate the effect of GDC-0449 on the QT/QTc interval in healthy female subjects of non-childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Female, over 45 years of age
* In good health, as determined by the absence of clinically significant findings from the screening visit
* Body mass index between 18 and 32 kg/m^2 inclusive, with a body weight > 45 kg
* Of non-childbearing potential

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiac, vascular, endocrinological, hematological, or allergic disease; metabolic disorder; cancer; or cirrhosis
* Allergy to moxifloxacin or any quinolone antibiotics or any confirmed significant allergic reactions against any drug, or multiple allergies in the judgment of the investigator
* Personal or family history of congenital long QT syndrome or family history of sudden death
* Participation in an investigational drug or device study with an investigational drug within the last 3 months or six times the elimination half-life, whichever is longer, prior to Day 1 of the study

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-08-25 (Actual); Primary Completion 2011-03-18 (Actual); Study Completion 2011-03-18 (Actual)

PRIMARY OUTCOMES:
The QTcF (QT interval corrected by Fridericia's correction method) | Throughout study or until early discontinuation

SECONDARY OUTCOMES:
Change in ECG from baseline | Throughout study or until early discontinuation
Pharmacokinetic parameters of GDC-0449 | Throughout study or until early discontinuation
Incidence, nature and severity of adverse events | Throughout study or until early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jean Ayache, M.D., Study Director — Hoffmann-La Roche